CLINICAL TRIAL: NCT04444882
Title: Complications After Lumpectomy, Sentinel Node and Radiotherapy in Breast Cancer Patients and Physiotherapy Care
Acronym: COTUKI
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.120; 2020-A00966-33 (Other: ID RCB)
Record Dates: First submitted 2020-05-28; First posted 2020-06-24 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Breast Neoplasm
Keywords: postoperative complications; physiotherapy; rehabilitation; lumpectomy; sentinel node; radiotherapy
MeSH Terms: conditions — Breast Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To make an inventory of the physiotherapeutic care and the post-operative complications of patients who have undergone lumpectomy, sentinel node and radiotherapy treatment.

The investigators expect to see a lack of consultation of physiotherapists by patients despite a significant number of complications, impacting the quality of life.

DETAILED DESCRIPTION:
This study is observational and descriptive. For this purpose, patients meeting the inclusion and non-inclusion criteria can answer, if they wish, to an online questionnaire after having read the information and non-opposition letter.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer Patients
* Patients with a good command of French in order to understand the letter of information and the questionnaire.
* Patients treated at the "Couple Enfant Hospital" in Grenoble. We have chosen to take patients who have been operated on at least 3 months ago (average time of end of radiotherapy).

Exclusion Criteria:

* Patient having undergone a mastectomy or chemotherapy
* Patient with difficulties understanding, expressing or reading the French language
* Vulnerable patient or patient with impaired cognitive capacities (dementia, confusion)
* Patient subject to a legal protection measure or out of state to express her opposition (guardianship, curatorship)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study involves breast cancer patients who have undergone the following treatment: lumpectomy, sentinel node and radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Inventory of the physiotherapeutic care of patients who have undergone lumpectomy, sentinel node and radiotherapy treatment | 10 minutes
  Answers to the questionnaire part 2 "physiotherapy care". Questions 17, 18, 19, 20, 21, 22, 24, 25, 26. (étude descriptive)

SECONDARY OUTCOMES:
Description of the post-operative complications of patients who have undergone lumpectomy, sentinel node and radiotherapy treatment | 10 minutes
  Answers to the questionnaire part 2 " post-operative complications " Questions 16, 23, 27, 28.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Bordin-Goffin, Study Director — IFMK Saint Martin d'Hères
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No